CLINICAL TRIAL: NCT06854497
Title: The Impact of Non-motor Symptom on the Outcome of Stroke Patients: A Prospective Observational
Brief Title: The Impact of Non-motor Symptom on the Outcome of Stroke Subjects
Acronym: NMCHYIS
Status: Active, not recruiting | Type: Observational
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CYCH2765041; R112-03 (Other Grant/Funding Number: Ditmanson Medical Foundation Chiayi Christian Hospital, Chiayi City, Taiwan)
Record Dates: First submitted 2024-09-05; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Delirium; Fatigue; Depression; Insomnia; Sleep Apnea Syndrome (OSAS); Skin Lesion; Dementia
Keywords: skin lesion; stroke; delirium; fatigue; sleep disorder; depression; outcomes
MeSH Terms: conditions — Delirium; Fatigue; Depression; Sleep Initiation and Maintenance Disorders; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Dementia; Stroke; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: MMSE (Mini-Mental State Examination),NIHSS (NIH Stroke Scale) and mRS (Mordified Rankin Score), Confusion Assessment Methods (CAM), PSQI Pittsburgh Sleep Quality Index, Respiratory polygraphy — Respiratory polygraphy will be performed during acute stroke period, to evaluate the relationship between sleep apnea and stroke evolution.

SUMMARY:
The most common symptoms of stroke were focal weakness, hemiparesis, speech disturbance, diplopia and ataxia. Beside those symptoms, there are still many symptoms occurring after stroke, which may affect the life quality of participants. Compared to motor symptoms, the study of these non-motor symptoms was too small.

At present, the most reported non-motor symptoms after stroke are sleep disorder, depression and post-stroke pain. There are still many symptoms that were not investigated.

The study investigates the prevalence of non-motor syndromes in acute ischemic stroke patients and the impact of these syndromes on the outcome of ischemic stroke patients. The non-motor syndromes that were researched include dizziness, pain, skin lesions, sensory impairment, fever, infection, delirium, depression, insomnia, confusion, delirium and headache.

Delirium may occur after stroke. Delirium may impair the mentality, thinking, attention and consciousness level of participants. There are many causes reported attributed to confusion including infection, old age, stroke, hemorrhage… Early diagnosis and early treatment for confusion may improve outcome and decrease mortality in stroke populations. One of the aims of the study is to investigate the prevalence, causes and outcome of treatment in stroke populations who hospitalized to the hospital. Fatigue is a feeling of tiredness or lack of energy. Fatigue is not the same as the feeling drowsy or sleepy. When a person is fatigued, they lose motivation and energy. Fatigue may be mild to severe. It may be related to a physical or mental health condition. The study investigates the prevalence and impact of fatigue on stroke populations' outcomes. In depression, a person experiences a loss of pleasure or interest in activities and feels sad, irritable, and empty. Post-stroke depression is common. When a stroke person has a depressed mood, they may have no motivation for activity. This may interfere with physical therapy and affect the outcome of a stroke. The study investigates post-stroke depression prevalence and impact. The study investigates the prevalence and impact of sleep apnea on stroke outcome.

DETAILED DESCRIPTION:
Delirium may occur after stroke. Delirium may impair the mentality, thinking, attention and consciousness level of participants. There are many causes reported attributed to confusion including infection, old age, stroke, hemorrhage… Early diagnosis and early treatment for confusion may improve outcome and decrease mortality in stroke populations. One of the aims of the study is to investigate the prevalence, causes and outcome of treatment in stroke populations who undergo hospitalization to the hospital. Fatigue is a feeling of tiredness or lack of energy. Fatigue is not the same as being drowsy or sleepy. When a person is fatigued, they lose motivation and energy. Fatigue may be mild to severe. It may be related to a physical or mental health condition. The aim of the study is to investigate the prevalence and impact of fatigue on the outcome of stroke populations. Depression is a person experiencing depressed mood (saddy, irritable, and empty) or loss of pleasure or interest in activities. Post-stroke depression is common. When a stroke person has a depressed mood, they lose motivation in activity which may interfere with physical therapy and affect stroke outcomes. The study explores the prevalence and impact of post-stroke depression.

Methods The study included all potentially participants who were referred to the hospital with a stroke. Exclusion criteria: 1. Age less than 20 years. 2. Severe dementia (MMSE lower than 10. 3. No agree to participate in the study.

All participants were followed-up for 3 months after stroke onset. During the acute ischemic stroke stage, researchers will evaluate participants' skin, ask participants about symptoms of headache, pain, dizziness, sensory complaint, sleep condition, evaluate participants' emotion condition everyday till discharge and follow up till 3 months after stroke onset. The study also researches the impact of non-motor syndromes on stroke outcomes.

The scales used to evaluate non-motor syndromes were listed.

Delirium study: Confusion Assessment Methods (CAM) is used to evaluate the consciousness of participants admitted to ICU, Brief Confusion Assessment Methods (bCAM) is used to evaluate the consciousness of participants who are not admitted to ICU.

DSM-V diagnosis criteria of confusion were used to diagnose confusion. The time of confusion evaluation is every day in the first week after stroke onset. Investigator also evaluates MMSE, NIHSS, mRS.

Fatigue study Fatigue severity Index was used to evaluate fatigue severity. Fatigue was evaluated in the first week, and 3 months after the stroke. Investigator also evaluates MMSE, NIHSS, mRS.

Post-stroke depression study Beck Depression Inventory and Hospital anxiety and depression Scale were used to evaluate the mood of the participants. Participants' mood was evaluated in the first week, and 3 months after stroke onset. Investigator also evaluates MMSE, NIHSS and mRS. MMSE was evaluated on the first day of admission. NIHSS was evaluated on the first day of admission and discharge. mRS was evaluated at day of discharge, and 3 months. The Berlin Questionnaire was used to evaluate the risk of sleep apnea. Respiratory polygraphy was used to evaluate sleep apnea during admission.

Description of the scale were used in the study A. Confusion Assessment Methods (CAM)

CAM is based on four key diagnostic features:

1. Acute Onset and Fluctuating Course - The sudden development of confusion with variations in severity over time.
2. Inattention - Difficulty focusing or maintaining attention.
3. Disorganized Thinking - Illogical or incoherent thoughts.
4. Altered Level of Consciousness - A state of hyper alertness or lethargy. For a positive delirium diagnosis, participant needs present with first two features along with either the third or fourth.

B. Mini-Mental State Examination (MMSE) MMSE

1. MMSE consists of 30 questions divided into five cognitive domains, Include orientation, registration, attention and calculation, recall, language and praxis.
2. 24 - 30: Normal cognitive function, 18 - 23: Mild cognitive impairment 10 - 17: Moderate cognitive impairment, 0 - 9: Severe cognitive impairment.

C. National Institutes of Health Stroke Scale (NIHSS)

1. NIHSS consists of 11 components, total score range from 0 to 42.
2. 0: No stroke, 1-4: Minor stroke, 5-15: Mo derate stroke, 15-20: Moderate/severe stroke, 21-42: Severe stroke

D. Modified Rankin Score The score of 0-3 indicates mild to moderate disability. Score of 4-5 indicates severe disability. 6 indicates death.

E. Berlin Questionnaire The Berlin Questionnaire consists of 10 questions divided into three categories. According to the response, participants were classified as high risk or low risk of obstructive sleep apnea.

F. Fatigue Severity Scale (FSS) The FSS questionnaire contains nine statements. Participants read each statement and circle a number from 1 to 7. FSS score over 36 is considered to have fatigue.

G. Apnea-hypopnea index (AHI) Respiratory polygraphy was used to evaluate sleep apnea within the first Week after stroke onset. AHI over 15 is considered as sleep apnea.

H. 36-Item Short Form Health Survey (SF-36) SF-36 is used to evaluate quality of life.

SF-36 consists of 36 questions that assess eight health domains:

1. Physical Functioning (PF) - Measures limitations in performing physical activities (e.g., walking, climbing stairs).
2. Role Physical (RP) - Assesses role limitations due to physical health problems.
3. Bodily Pain (BP) - Evaluates the impact of pain on daily activities.
4. General Health (GH) - Measures overall personal health perceptions.
5. Vitality (VT) - Assesses energy levels and fatigue.
6. Social Functioning (SF) - Evaluates the impact of health on social activities.
7. Role Emotional (RE) - Measures role limitations due to emotional problems.
8. Mental Health (MH) - Assesses psychological well-being and distress. Each domain is scored on a 0 to 100 scale, where higher scores indicate Better health status.

Outcome measure Primary outcome Functional outcome Modified Rankin Score (mRS) is used to evaluate the functional outcome of the participants up to 3 months after stroke onset.

The mRS score (0 to 6), scores of 0-3 indicate mild to moderate disability. a score of 4-5 indicates severe disability, and 6 indicates death. In the study, a mRS over 2 is considered poor outcome.

Secondary outcome Quality of life 36-Item Short Form Health Survey (SF-36) used to evaluate quality of life for 3 months. SF-36 consists of 36 questions that assess eight health domains. Each domain is scored on a 0 to 100 scale, where higher scores indicate better health status.

A score lower than 60 in a domain is considered as low quality in the health domain..

ELIGIBILITY:
Inclusion Criteria:

* 1. Acute stroke within 1 week.
* 2. Ischemic stroke was confirmed by magnetic resonance imaging.

Exclusion Criteria:

* 1. Patient not agree the study.
* 2. Patient cannot communication.
* 3. Severe dementia (mmse <10)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients admitted to hospital within 1 week of stroke onset. Brain magnetic resonance inaging confirmed ischemic. Patient age between 20 and 90 years old were included the study. Exclusion criteria were 1. patient older than 90 years old. 2. patient cannot communication included severe dementia, aphasia and consciousness disturbance. 3. Patient do not agree participate the study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | Participants are followed-up up to 3 months after stroke onset.
  Modified Rankin Score (mRS) is used to evaluate the functional outcome of the participants up to 3 months after stroke onset.
  The mRS score (0 to 6), scores of 0-3 indicate mild to moderate disability. a score of 4-5 indicates severe disability, and 6 indicates death. In the study, a mRS over 2 is considered poor outcome.

SECONDARY OUTCOMES:
Quality of life in ischemic stroke patients | follow patient daily activity of life at 3 month after stroke
  Quality of life 36-Item Short Form Health Survey (SF-36) used to evaluate quality of life for 3 months. SF-36 consists of 36 questions that assess eight health domains. Each domain is scored on a 0 to 100 scale, where higher scores indicate better health status. A score lower than 60 in a domain is considered as low quality in the health domain.

CONTACTS AND LOCATIONS:
Overall Officials: Cheung-Ter Ong, Master, Principal Investigator — Ditmanson Medical Foundation Chiayi Christian Hospital Neurologist
Locations (1):
- Ditmanson Medical Foundation Chiayi Christian Hospital, Chiayi City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No